CLINICAL TRIAL: NCT05140811
Title: Phase 1/Phase 2 Study of IMM01 Combined With Azacitidine in Patients With AML and MDS
Brief Title: A Study of IMM01 Combined With Azacitidine in Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Collaborators: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMM01-02
Record Dates: First submitted 2021-10-17; First posted 2021-12-01 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Relapse/Refractory AML (Experimental): IMM01 and Azacitidine in Relapse/Refractory AML
  Interventions:
  Drug: IMM01 Drug: Azacitidine
  Interventions: Drug: IMM01; Drug: Azacitidine
- Relapsed or Refractory MDS (Experimental): IMM01 and Azacitidine in Relapse/Refractory MDS
  Interventions:
  Drug: IMM01 Drug: Azacitidine
  Interventions: Drug: IMM01; Drug: Azacitidine
- Treatment naive AML (Experimental): IMM01 and Azacitidine in treatment naive AML
  Interventions:
  Drug: IMM01 Drug: Azacitidine
  Interventions: Drug: IMM01; Drug: Azacitidine
- Treatment naive MDS and naive CMML (Experimental): IMM01 and Azacitidine in treatment naive MDS and naive CMML
  Interventions:
  Drug: IMM01 Drug: Azacitidine
  Interventions: Drug: IMM01; Drug: Azacitidine

INTERVENTIONS:
Drug: IMM01 — IMM01 is intravenously once a week, every 28 days for a treatment cycle;
  Other Names: IMM01 Ingection
Drug: Azacitidine — Azacitidine 75 mg/m/ day is administered subcutaneously for 7 consecutive days, with each 28-day treatment cycle planned for 6 treatment cycles
  Other Names: Vidaza

SUMMARY:
This trial is an open-lable , multi-center, Phase 1/Phase 2 study that will evaluate the safety, tolerability, Pharmacokinetics, Pharmacodynamics and and immunogenicity of IMM01 combined with Azacitidine in patients with Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS).

DETAILED DESCRIPTION:
Main study purpose:

* To evaluate the safety and tolerability of IMM01 combined with Azacitidine in patients with AML and MDS.
* To explore the Maximum Tolerated Dose (MTD) of IMM01 combined with Azacitidine, and determine the phase 2 clinical recommended dose (RP2D) of IMM01 combined with Azacitidine.

Secondary study purpose:

* To evaluate the efficacy of IMM01 combined with Azacitidine in patients with AML and MDS.
* To evaluate the Pharmacokinetics and Pharmacodynamics of IMM01 combined with Azacitidine, in patients with AML and MDS.

Exploratory study purpose:

• To evaluate the immunogenicity of IMM01 combined with Azacitidine in patients with AML and MDS.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent.
2. Males and females ≥18 years of age
3. The Eastern Oncology Collaboration (ECOG) Status of ≤2
4. Life expectancy of at least 3 months.
5. Women and men of reproductive age must agree and use effective contraception during the study period and for three months after the last administration of IMM01, and women of reproductive age must have negative pregnancy test results within seven days prior to administration.
6. White blood cell count ≤ 20×10⁹/L before the first treatment of the study drug (treatment with hydroxyurea is permitted, but not within 3 days before the first treatment of the study drug).
7. Bone marrow aspiration and bone marrow biopsy were agreed during screening and treatment.
8. For those who have received previous chemotherapy or targeted drug therapy, the interval between the first drug administration should be more than 2 weeks;Prior treatment with chimeric antigen receptor T cells (CAR T cells) should be discontinued for at least 12 weeks after initial dosing(for Cohort 1 and 2).
9. Non-hematological adverse reactions have been restored to grade 1 and below (NCI-CTC AE v5.0, except residual hair loss effect),in patients with previous chemotherapy and targeted drug therapy. Hematologic adverse reactions recovered to investigatory-determined acceptance of study drug administration (for cohort 1 and 2).
10. Appropriate organ functions.

Exclusion Criteria:

1. Received anti-CD47 antibody or SIRPα fusion protein research drugs.
2. Who has received allogeneic hematopoietic stem cell transplantation and other organ transplants; Autologous hematopoietic stem cell transplantation less than six months.
3. Central nervous system leukemia orcentral nervous system invasion.
4. Developed other malignant tumors within 5 years prior to enrollment.Except:

   Cured carcinoma in situ and non-melanoma skin cancer of the cervix; Complete remission of disease at least 2 years prior to initial administration and no need for antineoplastic therapy.
5. Patients with a history of active autoimmune diseases;
6. Major surgery within 4 weeks prior to initial treatment;
7. Subjects requiring systemic corticosteroids (equivalent to >10 mg prednisone/day) or other immunosuppressive agents within 14 days prior to initial treatment or during the study period;
8. Hypertension (systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg) or pulmonary hypertension or unstable angina that is also not controlled by medication;
9. Patients with a history of arterial or deep vein thrombosis within the 6 months prior to enrollment, or evidence or history of bleeding tendency within the 2 months prior to enrollment, regardless of severity.
10. Severe gastrointestinal diseases;
11. With acute lung disease, pulmonary fibrosis, Severe dyspnea, lung insufficiency or continuous oxygen inhalation.
12. Patients who have been severely infected within 4 weeks prior to initial administration;
13. Active hepatitis B or hepatitis C ; human immunodeficiency virus (HIV) antibody is positive.
14. Live attenuated vaccine should be administered within 4 weeks prior to initial administration.
15. Patients with a history of severe allergy to protein drugs (CTCAE V5.0 grade > 3); Or the patient is allergic to azacytidine.
16. Participate in clinical trials of other drugs 28 days prior to initial dosing.
17. A history of prior neurological or mental disorders, such as epilepsy, dementia, or alcohol, drug or substance abuse, affects compliance.
18. Other conditions that the investigator considers inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-02-05 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate and the grade (severity) of dose-limiting toxicities (DLTs) of IMM01 combination azacitidine | Though end of DLT evaluation period,up to approximately 28 days.
  To be summarized using descriptive statistics
Maximum Tolerated Dose (MTD) | Dose-limiting toxicities will be evaluated during the first cycle (28 days) of treatment.
  MTD is the highest dose in patients with DLT incidence <1/3.For a dose group to be assessed as MTD, at least 6 DLT data must be available to evaluate the subject.

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax | Within 60 minutes prior to infusion on Cycle 1 Day 1, Day 8, Day 15 and Cycle 2-6 Day 1 (28 days cycle).10 minutes post-infusion on Cycle 1 Day 15 and Cycle 6 Day 22 (28 days cycle ) .10 minutes and 4 hours post-infusion on Cycle 1 Day 1 (28 days cycle).
  Maximum observed concentration in serum
Pharmacokinetics - AUC | Within 60 minutes prior to infusion on Cycle 1 Day 1, Day 8, Day 15 and Cycle 2-6 Day 1 (28 days cycle).10 minutes post-infusion on Cycle 1 Day 15 and Cycle 6 Day 22 (28 days cycle ) .10 minutes and 4 hours post-infusion on Cycle 1 Day 1 (28 days cycle).
  Area under the serum concentration - time curve
Pharmacokinetics - tmax | Within 60 minutes prior to infusion on Cycle 1 Day 1, Day 8, Day 15 and Cycle 2-6 Day 1 (28 days cycle).10 minutes post-infusion on Cycle 1 Day 15 and Cycle 6 Day 22 (28 days cycle ) .10 minutes and 4 hours post-infusion on Cycle 1 Day 1 (28 days cycle).
  Time to peak (maximum) serum concentration
Pharmacokinetics - T1/2 | Within 60 minutes prior to infusion on Cycle 1 Day 1, Day 8, Day 15 and Cycle 2-6 Day 1 (28 days cycle).10 minutes post-infusion on Cycle 1 Day 15 and Cycle 6 Day 22 (28 days cycle ) .10 minutes and 4 hours post-infusion on Cycle 1 Day 1 (28 days cycle).
  Terminal half-life (T1/2)
Response Rate | When the last subject enrolled completes approximately 12 months of treatment
  Response determined per European LeukemiaNet response criteria:
  CR = bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count > 1.0 x 10e9/L; platelet count > 100 x 10e9/L; and independence of red cell transfusions.
  CRi = all CR criteria except for residual neutropenia (< 1.0 x 10e9/L) or thrombocytopenia (< 100 x 10e9/L)].
  To evaluate clinical benefit defined as CR, CRi, morphologic leukemia-free state, and partial remission (PR).
Overall Remission (OR): | When the last subject enrolled completes approximately 12 months of treatment
  Response Criteria are according to the Modified IWG (International Working Group) Response Criteria in Myelodysplasia.CR: bone marrow evaluation shows less than or equal to (<=) 5% blasts; normal maturation of all cells lines (mCR), peripheral blood evaluation shows hemoglobin >= 11 gram per deciliter (g/dL), neutrophils >= 1000/mL, platelets >= 100,000/mL, 0% blasts; PR: Same as CR, except blasts decrease by >=50%, still greater than 5% in bone marrow. Hematologic improvement are measured in participants with pretreatment abnormal values: hemoglobin level less than 110 g/L (11 g/dL) or red blood count (RBC)-transfusion dependence, platelet count <100 x 10^9/L or platelet-transfusion dependence, absolute neutrophil count (ANC) less than 1.0 x 10^9/L.

OTHER OUTCOMES:
Exploratory Endpoint | In cycle 1(each cycle is 28 days) and cycle 4, 6, 8, 10, and 12, at the end of treatment or early study withdrawal, and 30 days after the last dose.
  Anti-drug Antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Beijing gobroad boren hospital, Beijing
  - Peking university third hospital, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - Chongqing university cancer hospital, Chongqing
  - Second Affliated Hospital of Army Medical University, Chongqing
  - Fujian medical university union hospital, Fuzhou
  - Ganzhou People's Hospital, Ganzhou
  - Guangdong provincial people hospital, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Zhujiang Hospital, Southern Medical University/The Second School of Clinical Medicine, Southern Medical University, Guangzhou
  - The first affiliated hospital zhejiang university school of medicine, Hangzhou
  - The first affiliated hospital of nanchang University, Nanchang
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai sixth's hospital, Shanghai
  - Tongren hospital shanghai jiaotong university school of medicine, Shanghai
  - Shengjing Hospital Affiliated to China Medical University, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - Tianjin Blood Disease Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The affiliated hospital of Xuzhou medical university, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
  - The first affiliated hospital of Zhengzhou University, Zhengzhou